CLINICAL TRIAL: NCT04420143
Title: An Assessment of the Safety and Performance of the MLX® Medial Lateral and XLX ACR® Expandable Lumbar Interbody Implants for the Treatment of Patients With Degenerative Conditions of the Thoracic and/or Lumbar Spine
Brief Title: MLX/XLX ACR Expandable Lumbar Interbody Implants
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.EXP0120
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Degenerative Scoliosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- MLX - Medial Lateral Expandable Lumbar Interbody System: Patients who underwent lumbar interbody fusion with the MLX expandable interbody implant will be included in the MLX - Medial Lateral Expandable Lumbar Interbody System cohort.
- XLX ACR Interbody System: Patients who underwent lumbar interbody fusion with the XLX ACR expandable interbody implant will be included in the XLX ACR Interbody System cohort.

SUMMARY:
The objective of this study is to evaluate the safety and performance of thoracic and/or lumbar spine surgery using the MLX and XLX ACR interbody implants as measured by reported complications, radiographic outcomes, and clinical patient outcomes. This study is being undertaken to identify possible residual risks and to clarify mid- to long-term clinical performance that may affect the benefit/risk ratios of the MLX and XLX ACR interbody implants.

DETAILED DESCRIPTION:
Patients considered for this study will have previously undergone surgery for their spinal condition according to the standard of care of the practitioner. All patients at a given site with surgeries that meet eligibility requirements will be included in the study and available progress notes, medical records, patient-reported outcomes (PROs), radiographs, and complications will be obtained from the medical records.

The safety and performance of the MLX and XLX ACR interbody implants will be assessed using the following:

1. Complications attributable to the use of the associated interbody implant as noted in surgical summaries, progress notes, and hospital records
2. Neurologic status, symptoms, and subject self-reported clinical outcomes (e.g., pain and disability), as available
3. Radiographic outcome (fusion) and description of device status from plain film radiographs and computed tomography (CT) scan(s), as available

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were ≥18 years of age at the time of surgery
2. Underwent spine surgery using either MLX or XLX ACR interbody implant (NuVasive, Inc., San Diego, CA) at:

   1. One or two adjacent thoracic and/or lumbar levels for degenerative disc disease or degenerative spondylolisthesis, or
   2. Any number of thoracic and/or lumbar levels for degenerative scoliosis (defined as >10º coronal curve)
3. Interbody fusion with autograft and/or allograft (i.e., cancellous and/or corticocancellous allograft bone)
4. NuVasive supplemental internal fixation cleared by the applicable regulatory body for use in the thoracolumbar spine

Exclusion Criteria:

1. Use of any bone graft with the associated interbody implant that is not FDA-cleared for use within interbody implants.

   Examples of these include:
   1. Bone morphogenetic protein (BMP) (e.g., Infuse (Medtronic))
   2. Synthetic bone graft extenders (e.g., AttraX (NuVasive), Formagraft (NuVasive), Mastergraft (Medtronic), Vitoss (Stryker), Actifuse (Baxter), nanOss (RTI Surgical), Fibergraft (Prosidyan/Depuy Synthes), ChronOs (Depuy Synthes))
   3. Demineralized bone matrices (DBM) regulated as medical devices by the FDA (e.g., Grafton Putty/Gel (Medtronic), DBX (MTF/Depuy Synthes), Accell Evo3 (IsoTis), Propel Putty/Gel (NuVasive))
   4. Peptide enhanced bone graft (e.g., iFactor (Cerapedics))
2. Previous lumbar fusion surgery at the currently treated level(s) (adjacent-level surgery is acceptable)
3. Systemic or local infection (latent or active) or signs of local inflammation documented at the time of surgery
4. Patient was involved in active litigation relating to the spine during the surgical/postoperative period (worker's compensation claim is allowed if it is not contested)
5. Inadequate bone stock or bone quality documented at the time of surgery
6. Known sensitivity to materials implanted documented at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 90 (75 MLX, 15 XLX ACR) subjects will be enrolled in this multicenter study by at least four investigative sites. A site may have more than one surgeon investigator contributing to the total site enrollment. As a retrospective study, enrollment goals will be determined with the surgeon investigator during site selection by the Sponsor and will be based on available case volume. The site will identify potential subjects who are more than three months from the surgery postoperative time point during the study duration for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Rate of Complications | At least three months
  Rate of complications (i.e., safety) attributable to use of the associated interbody implants (MLX or XLX ACR)
Proportion of Subjects with Improvement in Neurological Symptoms | At least three months
  The rate of improvement as compared to baseline in preoperative neurological symptoms will be measured using a standard motor/sensory neurological exam.

SECONDARY OUTCOMES:
Proportion of Subjects with Apparent Radiographic Fusion | 12 months or greater
  Proportion of subjects with apparent radiographic fusion at 12 months or greater postoperative, as imaging is available

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (4):
- United States (4):
  - Orthopaedic Specialty Institute, Orange, California
  - Lyerly Neurosurgery, Jacksonville, Florida
  - Carolina NeuroSurgery & Spine Associates, Charlotte, North Carolina
  - OrthoCarolina Research Institute, Charlotte, North Carolina